CLINICAL TRIAL: NCT01866774
Title: Evaluation of Fecal Calprotectin Screening and a Gastroenterology Questionnaire for Triaging Children With Chronic Abdominal Pain and/or Diarrhea Referred to a Pediatric Gastroenterology Service - A Randomized, Controlled Trial
Brief Title: Evaluation of Fecal Calprotectin Screening and a Gastroenterology Questionnaire for Triaging Children With Chronic Abdominal Pain and/or Diarrhea Referred to a Pediatric Gastroenterology Service
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary Investigator (AJN) left institution
Sponsor: Queen's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Q4415
Record Dates: First submitted 2013-01-03; First posted 2013-05-31 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Abdominal Pain; Chronic Diarrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fecal calprotectin level (Experimental): Fecal calprotectin level
  Interventions: Other: Fecal calprotectin level
- Symptom questionnaire (No Intervention)

INTERVENTIONS:
Other: Fecal calprotectin level
  Arms: Fecal calprotectin level

SUMMARY:
Triaging new pediatric gastroenterology consultations is challenging as both inflammatory and non-inflammatory gastrointestinal (GI) diseases can present with non-specific chronic abdominal pain and/or diarrhea. Examples of inflammatory GI diseases include Crohn's disease, ulcerative colitis and celiac disease and non-inflammatory GI diseases lactose intolerance, irritable bowel syndrome and non-ulcer dyspepsia. Inflammatory GI diseases require different investigations and treatment than non-inflammatory GI diseases and ideally, would be identified early. Higher priority triage of these patients would allow timely organization of further investigations including pertinent laboratory testing, radiologic studies and gastrointestinal endoscopies. These more invasive procedures are not needed in most patients presenting with non-specific gastrointestinal symptoms. Therefore, the investigators do not routinely ask for screening laboratory testing or other studies in children referred to our clinic.

Non-invasive screening tests for GI disorders may aid in appropriately triaging new consultations to pediatric gastroenterology. Calprotectin is a protein found in inflammatory cells called neutrophils. The concentration of calprotectin in stool reflects the presence of an inflammatory process occurring in the GI tract. Thus, testing for calprotectin has been proposed as a potentially useful test for detecting some inflammatory GI diseases, most notably Crohn's disease and ulcerative colitis. Alternatively, a simple gastrointestinal questionnaire of "red flag" symptoms and family history of GI disorders may also be of benefit. The investigators hypothesize that the use of fecal calprotectin and a screening GI questionnaire will aid in identifying children at higher risk of an inflammatory GI disorder. Subsequently, higher priority triaging of these patients will decrease the time to diagnosis of inflammatory GI disease.

This will be a single centre, stratified, randomized clinical trial conducted in Kingston, Ontario, Canada. Patients referred to the pediatric gastroenterology service without a known diagnosis for non-specific chronic abdominal pain and/or diarrhea will be asked to participate in the study. All patients who meet the inclusion criteria will be consented by telephone with a standard form. Consenting patients will be mailed the GI questionnaire and the fecal calprotectin test kit. The fecal calprotectin test kid includes instructions, a stool collection kit and return postage. All patients will be given the next available appointment with a pediatric gastroenterologist. Patients will then be randomized to receive either usual care (50%, 40 patients) or to have a screening fecal calprotectin (FC) measurement (50%, 40 patients). Patients in the FC group will have FC measured by the Quantum Blue® Rapid Calprotectin Assay. If the calprotectin level is high (above 50 μg/g), the patient will be contacted again by telephone and given a new appointment time (within 14 working days). This study may have a positive impact by demonstrating a novel method for decreasing the time to diagnosis of inflammatory GI disease.

ELIGIBILITY:
Inclusion criteria:

* have been referred to the pediatric gastroenterology service at the Kingston University Hospital Network for abdominal pain or chronic diarrhea
* be between 5 to 17 years of age

Exclusion criteria:

* overt signs and symptoms of an inflammatory gastrointestinal disease in the referral letter (will triaged with high priority within 14 working days
* evidence of GI bleeding, extraintestinal manifestations of inflammatory bowel disease, significant weight loss or laboratory abnormalities

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2013-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Time to final diagnosis | Up to 12 months from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Angela Noble, MD, Principal Investigator — Kingston Health Sciences Centre
Locations (2):
- Canada (2):
  - Kingston University Hospital Network, Kingston, Ontario
  - Queen's University, Kingston, Ontario